CLINICAL TRIAL: NCT02278042
Title: A Comparison of the Neurocognitive and Metabolic Effects of Fructose, Glucose, High Fructose Corn Syrup and Sucrose at Normal Population Consumed Levels in Adults Ages 20-60 Years Old
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rippe Lifestyle Institute (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 20131024
Record Dates: First submitted 2014-10-27; First posted 2014-10-29 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Conditions: None. Focus: Understanding the Obesogenic Potential of Fructose Containing Sugars

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 9% Fuctose (Active Comparator): Milk Sweetened with fructose in an amount that the added fructose contributes 9% of the calories required for weight maintenance.
  Interventions: Other: Beverage Consumption
- 18% Sucrose (Active Comparator): Milk Sweetened with sucrose in an amount that the added sucrose contributes 18% of the calories required for weight maintenance.
  Interventions: Other: Beverage Consumption
- 18% High fructose corn syrup (Active Comparator): Milk Sweetened with High fructose corn syrup (HFCS) in an amount that the added HFCS contributes 18% of the calories required for weight maintenance.
  Interventions: Other: Beverage Consumption
- 9% Glucose (Active Comparator): Milk Sweetened with glucose in an amount that the added glucose contributes 9% of the calories required for weight maintenance.
  Interventions: Other: Beverage Consumption
- Unsweetened Milk (Active Comparator): Unsweetened milk consumed in amount the contributes 18% of the calories required for weight maintenance.
  Interventions: Other: Beverage Consumption

INTERVENTIONS:
Other: Beverage Consumption

SUMMARY:
The purpose of this study is to investigate the acute and chronic effects of consumption fructose containing sugars and glucose in a real word setting when consumed in a manner and amount typical in the American diet.

DETAILED DESCRIPTION:
Detailed description (Why and How?) Fructose is known to be metabolized differently than the other common monosaccharides. In addition to the well know lipogenic effects, more recent evidence has shown that the acute changes in hormones and metabolic parameters that control appetite and energy regulation when with fructose consumption may promote caloric overconsumption and, in the long-term, weight gain and deteriorations in insulin sensitivity. However, fructose is rarely consumed in isolation, but instead is consumed in combination with other sugars (with glucose in the case of the two most common sources of fructose: high fructose corn syrup (HFCS) and sucrose, or as part of a mixed macronutrient meal. As such, the practical significance of these short-term findings of isolated monosaccharide consumption is limited.

AIM 1: investigate the response to ten weeks of daily consumption of typical levels of different fructose containing sugars and glucose on measures of glucose and insulin metabolism.

AIM 2: To investigate whether ten weeks of daily consumption changes the fat content of the liver, skeletal muscles or abdomen.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the ages of 20-60 years of age.
* Body Mass Index (BMI) 21.0 - 35.0

Exclusion Criteria:

* More than a 3 percent change in weight within the 3 months prior to enrollment in the study.
* History of thyroid disease, but not taking medication or medication dosage changed one or more times over last 6 months. History of thyroid disease and on a stable dose of prescription medication for 6 months or longer is acceptable.
* Currently taking a prescription medication for weight loss. If subject is willing to discontinue prescription medication(s) immediately and willing to refrain from taking medication(s) for duration of study, he/she may be enrolled after a four-week washout period.
* Currently taking any over-the-counter weight loss supplement(s). If subject is willing to discontinue supplement(s) immediately and willing to refrain from taking supplement(s) for duration of study, he/she may be enrolled after a two-week washout period.
* Currently enrolled in commercial weight loss program (e.g. Jenny Craig, Weight Watchers) or self-help group (e.g. TOPS, Overeaters Anonymous). If subject is willing to discontinue program immediately and willing to refrain from program for duration of study, he/she may be included after a two-week washout period.
* Diagnosed with prediabetes or frank diabetes (Type I or Type II).
* History of major surgery within three months of enrollment.
* History of heart problems (e.g. angina, bypass surgery, MI, etc.) within three months prior to enrollment.
* Presence of implanted cardiac defibrillator or pacemaker.
* Uncontrolled hypertension/high blood pressure.
* History of a surgical procedure for weight loss at any time (e.g. gastroplasty, gastric by-pass, gastrectomy or partial gastrectomy).
* Gastrointestinal disorders including chronic malabsorptive conditions, peptic ulcer disease, Crohn's disease, chronic diarrhea or active gallbladder disease.
* History of inflammatory bowel disease
* History of fatty liver
* History or presence of cancer. Persons with successfully resected basal cell carcinoma of the skin may be enrolled if treatment completed more than 6 months prior to enrollment.
* History of clinically diagnosed eating disorders including anorexia nervosa, bulimia nervosa or binge eating disorder.
* Women who are pregnant, lactating or trying to become pregnant.
* Currently taking any prescription medication for less than 3 months.
* Currently consuming >14 alcoholic drinks (1 drink = 12 fl oz beer, 4 fl oz wine or 1.5 fl oz liquor) per week and/or unwilling to limit intake to less than 3 drinks per week during study participation.
* Known allergy to HFCS, sucrose, fructose or glucose.
* History of alcohol dependency
* Participation in another clinical trial within 30 days prior to enrollment.
* Lactose intolerance
* Currently smoking cigarettes
* Any clinically significant food allergy

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 225 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change in glucose tolerance | 10 weeks (Baseline and week 10)
  Change in glucose Area Under the Curve (AUC) in response to a standard 2 hour Oral Glucose Tolerance Test
Change in Insulin Sensitivity | 10 weeks (Baseline and week 10)
  Change in 1) insulin AUC in response to a standard 2 hour Oral Glucose and Matsuda Insulin Sensitivity Index

SECONDARY OUTCOMES:
Change in fat content of the liver | 10 weeks (baseline and Week 10)
  Change in fat content of the liver as determined by Magnetic Resonance Spectroscopy (MRS)
Change in fat content of the abdomen | 10 weeks (baseline and Week 10)
  Change in fat content of the abdomen as determined by MRS
Change in fat content of the skeletal muscles | 10 weeks (baseline and Week 10)
  Change in fat content of the Vastus Lateralis and Gluteus Maximum as determined by MRI.
Change in hypothalamic activity | 10 weeks (baseline and Week 10)
  Change in hypothalamic activity in response to consumption of test beverages consumed as part of a standardized, mixed nutrient meal will be measured by functional MRI. Changes from baseline (mean percent signal change) will be determined after 10 weeks of daily consumption of the test beverage as part of the usual diet

CONTACTS AND LOCATIONS:
Locations (1):
- Rippe Lifestyle Institute, Celebration, Florida, United States